CLINICAL TRIAL: NCT01378416
Title: A Phase I Pharmacokinetic Trial of Decitabine (Dacogen) Administered as a 3-hour Infusion to Patients With Acute Myelogenous Leukemia or Myelodysplastic Syndrome
Brief Title: Pharmacokinetic Trial of Decitabine (Dacogen) Administered as a 3-hour Infusion to Patients With Acute Myelogenous Leukemia or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Gerard Kennealey, MD, Eisai Medical Research Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DACO-018
Record Dates: First submitted 2008-09-30; First posted 2011-06-22 (Estimated); Results first posted 2011-06-22 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Leukemia
Keywords: Acute myelogenous leukemia; myelodysplastic Syndrome; cancer
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Neoplasms | interventions — Decitabine

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Decitabine (Dacogen)

INTERVENTIONS:
Drug: Decitabine (Dacogen) — Intravenous injection; total dose-per-cycle was 135 mg/m^2 of decitabine.
  Other Names: Dacogen

SUMMARY:
The purpose of this study is to determine the pharmacokinetics (PK) of decitabine administered to patients with myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

Each patient had to meet the following criteria to be eligible for the study:

1. Patients with MDS (de novo or secondary) must have been 60 years or older and have had disease fitting any of the recognized French-American-British classifications OR chronic myelomonocytic leukemia (with white blood cell [WBC] <12,000/μL) AND have had an International Prognostic Scoring System score of ≥1.5 as determined by complete blood count, bone marrow assessment and bone marrow cytogenetics within 30 days of study entry.
2. Patients with AML (≥30% bone marrow blasts) must have been age 18 years or older and had previously received standard induction chemotherapy and/or had failed approved therapies.
3. Must have had Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
4. Must have signed an Institutional Review Board (IRB)-approved informed consent form, indicating his/her awareness of the investigational nature of this study and its potential hazards prior to initiation of any study-specific procedures or treatment.
5. Must have had adequate renal and hepatic function (creatinine ≤2.0 mg/dL, total bilirubin <2.0 mg/dL, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <3.0 X institutional upper limit of normal).
6. Must have had life expectancy of at least 12 weeks.
7. Must have recovered from all toxic effects of all prior therapy before entry into this study.

Exclusion Criteria:

1. Patients with MDS must not have been candidates for high-dose chemotherapy, bone marrow or stem cell transplant.
2. Must not have had acute promyelocytic leukemia (M3 classification).
3. Must not have received immunosuppressive therapy for 30 days prior to study entry.
4. Must not have had central nervous system (CNS) leukemia.
5. Must not have received systemic corticosteroids, interferon, interleukins or other hormonal therapy within 30 days prior to study entry. Use of corticosteroids (topical and inhaled corticosteroids) was permitted and prophylactic steroids may have been used to treat or prevent transfusion reactions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-04; Primary Completion 2006-01 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Kennealey, MD, Study Director — Eisai Medical Research (formerly MGI Pharma Inc.)
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Decitabine: A 15 mg/m^2 dose was administered as a 3-hour IV infusion every 8 hours for 3 consecutive days in acute myelogenous leukemia/myelodysplastic syndrome patients.
Period: Overall Study
Arm/Group | Decitabine
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Decitabine
Number analyzed (Participants) | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 68.2 (11.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Secondary Outcome: Safety: The Most Frequently Reported Adverse Events (Regardless of Causality)
Description: Summary of All Adverse Events (AEs) by Maximum Grade Occurring in >= 10% Patients
Time Frame: 6 weeks
Measure: Number; unit: Participants
Arm/Group | Decitabine
Number analyzed (Participants) | 16
Participants
  Blood & Lymphatic System Disorders | 4
  Cardiac Disorders | 2
  Eye Disorders | 2
  Gastrointestinal Disorders | 11
  General Disorders & Administration Site Conditions | 14
  Infections and Infestations | 7
  Investigations - Weight decreased | 2
  Metabolism and Nutrition | 5
  Musculoskeletal and Connective Tissue Disorders | 6
  Nervous System Disorders | 8
  Psychiatric Disorders | 5
  Respiratory, Thoracic and Mediastinal Disorders | 13
  Skin and Subcutaneous Tissue Disorders | 9

2. Primary Outcome: Average Total Body Clearance (Calculated From Rate and Concentration)
Description: 3-hour IV infusion, every 8 hours for three consecutive days. Average Total Body Clearance was measured post first dose (Day 1), fourth dose (Day 2), and seventh dose (Day 3).
Time Frame: Day 1, Day 2, Day 3
Measure: Number; unit: L/hr/m^2
Arm/Group | Decitabine
Number analyzed (Participants) | 16
L/hr/m^2 | 129 (48.6)

3. Primary Outcome: Cmax (Maximum Plasma Concentration)
Description: 3-hour IV infusion, every 8 hours for three consecutive days. Cmax was measured post first dose (Day 1), fourth dose (Day 2), and seventh dose (Day 3).
Time Frame: Day 1, Day 2, Day 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Decitabine
Number analyzed (Participants) | 16
ng/mL
  Day 1 | 73.8 (48.6) [62.1 to 66]
  Day 2 | 64.8 (40.2) [54.5 to 62]
  Day 3 | 77.0 (62.5) [60.3 to 81.0]

4. Primary Outcome: Tmax (Time at Which Cmax First Observed)
Description: 3-hour IV infusion, every 8 hours for three consecutive days. Tmax was measured post first dose (Day 1), fourth dose (Day 2), and seventh dose (Day 3).
Time Frame: Day 1, Day 2, Day 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Decitabine
Number analyzed (Participants) | 16
hours
  Day 1 | 2.49 (0.70)
  Day 2 | 2.53 (0.69)
  Day 3 | 2.29 (0.63)

5. Primary Outcome: AUC (0-∞) - Area Under the Plasma Concentration-time Curve Extrapolated to Infinity
Description: 3-hour IV infusion, every 8 hours for three consecutive days. AUC (0-∞) was measured post first dose (Day 1), fourth dose (Day 2), and seventh dose (Day 3).
Time Frame: Day 1, Day 2, day 3
Measure: Mean (Standard Deviation); unit: ng∙hr/mL
Arm/Group | Decitabine
Number analyzed (Participants) | 16
ng∙hr/mL
  Day 1 | 163 (101)
  Day 2 | 152 (90.5)
  Day 3 | 158 (101)

ADVERSE EVENTS:
Arm/Group | Decitabine
Serious Adverse Events (participants affected / at risk) | 9/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Decitabine (N=16)
Febrile Neutropenia (Blood and lymphatic system disorders) | 3
Chills (General disorders) | 2
Disease Progression (General disorders) | 1
Pyrexia (General disorders) | 1
Bacteraemia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Sepsis (Infections and infestations) | 2
Acute Myeloid Leukemia Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral Ischemia (Nervous system disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Skin Necrosis (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Decitabine (N=16)
Palpitations (Cardiac disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Visual Accuity Reduced (Eye disorders) | 1
Visual Disturbance (Eye disorders) | 1
Abdominal Distention (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 2
Gingival Bleeding (Gastrointestinal disorders) | 2
Loose Tooth (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Proctalgia (Gastrointestinal disorders) | 1
Rectal Hemorrhage (Gastrointestinal disorders) | 1
Tongue Ulceration (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 2
Catheter Site Erythema (General disorders) | 1
Catheter Site Haematoma (General disorders) | 1
Catheter Site Related Reaction (General disorders) | 1
Chest Discomfort (General disorders) | 1
Chest Pain (General disorders) | 2
Chills (General disorders) | 4
Fatigue (General disorders) | 6
Feeling Hot (General disorders) | 1
Implant Site Bruising (General disorders) | 1
Implant Site Pain (General disorders) | 1
Oedema (General disorders) | 1
Pyrexia (General disorders) | 4
Thirst (General disorders) | 1
Graft Versus Host Disease in Liver (Immune system disorders) | 1
Bacteraemia (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Implant Site Cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Weight Decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 3
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 2
Cerebral Ischaemia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 1
Polyuria (Renal and urinary disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Painful Respiration (Respiratory, thoracic and mediastinal disorders) | 1
Paranasal Sinus Hypersecretion (Respiratory, thoracic and mediastinal disorders) | 2
Pharyngeal Erythema (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Blood Blister (Skin and subcutaneous tissue disorders) | 1
Drug Eruption (Skin and subcutaneous tissue disorders) | 1
Increased Tendency to Bruise (Skin and subcutaneous tissue disorders) | 1
Night Sweats (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin Necrosis (Skin and subcutaneous tissue disorders) | 1
Skin Nodule (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No